CLINICAL TRIAL: NCT02653404
Title: Observational Study to Compare IGRA and Mantoux Test in Children With Suspected Latent or Active TB Infection
Brief Title: IGRA and Mantoux Response in Children With Suspected Latent or Active TB Infection
Acronym: TBTubercolar
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, Francesca Montagnani, Dr., University of Siena
Other Study IDs: IGRAManPed2014
Record Dates: First submitted 2016-01-03; First posted 2016-01-12 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Tuberculosis, Pulmonary; Interferon-gamma Release Tests; Tuberculin Test
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cases: A blood sample necessary to perform QFT-GIT will be taken, together with other routine blood samples, from children with following diagnosis:
  * latent tuberculous infection: active TB contact, TST positive, lack of clinical and RX signs of active-TB
  * active TB: clinical and radiologic evidences of active-TB, positivity to microbial tests to BK
  * not infected: patients evaluated as TB contacts, with negative TST and negative clinical/radiological/microbial results for TB.
  Interventions: Other: IGRA test (QTF-GIT)

INTERVENTIONS:
Other: IGRA test (QTF-GIT) — blood sample for QFT-GIT will be taken together with other routine blood samples

SUMMARY:
The aim of this project is to analyze the potential contribution of IGRA test QuantiFERON-TB Gold In Tube test (QTF-GIT, Cellestis Limited, Carnegie, Victoria, Australia) in the diagnosis of tuberculosis (TB - active or latent) in pediatric subjects (0 and 17 year)s recently exposed to infection (indicated as "contacts") or with clinical suspicion of active TB, and to compare the results obtained with those of the TuberculinSkin Test (TST; gold standard). The project is expected to enroll up to 50 pediatric patients over a 4-year study. Children with access to Ambulatory structures or hospitalized at University Infectious Diseases Clinic or Pediatric Clinic, University Hospital of Siena, or with access to Ambulatory or hospitalized at Pediatric Clinic USL 9 Grosseto will be enrolled. Once obtained the informed consent of patients' parents or legal guardians, patients will be enrolled. The doctor will administer a clinical-anamnestic questionnaire, relative to the country of birth and residence, date of arrival in Italy and any stays in the country of origin (in case of foreign patient), travels abroad, risk factors for infectious diseases, type of contact with any index case, previous vaccination with BCG, date and outcome of the TST, clinical symptoms and signs suggestive of active TB, report of any instrumental investigation. Together with the collection of blood samples for routine purposes, an additional blood sample will be taken so to run IGRA test. Also patients for whom their medical doctor will independently order to run QTF-GIT test as necessary tool for the clinical diagnosis of TB will be included in the study.

A retrospective analysis will be performed on patient pertaining to participant Clinics, from 1 January 2012 to 31 May 2015. Such analysis will be performed on those patients for which their medical doctor requested both intradermal Mantoux and IGRA test.

Expected results:

* estimation of concordance between QuantiFERON-TB Gold In Tube and TST in pediatric patients exposed to TB, with or without latent TB infection
* Evaluation of the sensitivity of the test QTF-GIT in patients with active tuberculosis disease
* Evaluation of specificity of testQTF-GIT in not infected patients
* Evaluation on the possible use of QTF-GIT, together with TST, to improve the diagnosis of tuberculosis latent or active infection in pediatric subjects.
* Evaluation of the possible diagnostic use of QTF-GIT in the child <5 years.

DETAILED DESCRIPTION:
The diagnosis of tuberculosis in children is a complex procedure. The commonly used test is the tuberculin skin test (TST), which shows significant limitations such as cross-reactivity with the bacillus Calmette-Guerin (BCG) used for vaccination, and other environmental mycobacteria, the possible influence of age and the immunological status of the patient, the need to return to the hospital for the re-reading of the intradermal reaction. Since 2001, the Food and Drug Administration approved the first of a series of new tests, called Interferon-Gamma Release Assays (IGRAs), based on the release of interferon gamma by sensitized lymphocytes in the blood of the patient. Among them, the QuantiFERON-TBGold In Tube (QTF-GIT, Cellestis Limited, Carnegie, Victoria, Australia), is a highly specific test that measures, through an ELISA assay, the release of interferon-gamma production by lymphocytes in response to an antigenic challenge to Mycobacterium tuberculosis antigens. The antigens used in the test QTF-GIT (ESAT-6, CFP-10 and the sequence of TB7.7) are in fact absent from the vaccine strain BCG and in most nontuberculous mycobacteria, giving to the QTF-GIT test greater specificity than TST. Moreover, being an in vitro test, it does not require a return visit to the reading of the result (this is particularly important in screening of contacts), which is instead carried out in an instrument (and therefore objective) and, finally, thanks to the presence of an internal positive control, it is possible to evaluate the performance of tests and reduce possible technical errors. The QTF-GIT test gave significant results in adults in terms of sensitivity and specificity, as demonstrated by a large scientific literature, and is currently used in many hospitals, in combination with the TST, for the diagnosis of tuberculosis. Since September 2012, also the Siena University Hospital introduced the QTF-GIT assay as a diagnostic test for tuberculosis diagnosis in healthcare workers and in inpatient or outpatient tested positive TST requiring detailed diagnostic investigation (eg. Previous BCG vaccination, suspected atypical mycobacteriosis, eruptive events or other skin changes that contraindicate performing intradermal reaction).

Despite the important results obtained with the test QTF-GIT in adults, studies of specificity and sensitivity of the tests conducted in the pediatric age group are still limited. Some studies have shown a high specificity, while the sensitivity appears lower than the TST. The data are discordant, however, between the different studies, complicated by the fact that there is no real-Gold standard for the diagnosis of latent TB, and hence, further analysis is still needed.

While in adults the risk of progression from latent infection to active pulmonary disease is about 5-10%, in infants (<1 year old) this value increases up to about 30-40%, therefore the diagnosis and the treatment of latent infections is more than ever necessary to reduce the risk of developing the disease. Thus an urgent need to identify specific and sensitive diagnostic tools that would enable better diagnosis of TB in childhood, particularly in the age group under 5 years, as clearly expressed also by the European Centre for Disease Prevention and Control (ECDC) in guidelines "Use of Interferon-gamma release assays in support of TB diagnosis" and by the resolution of the Regional Council of Tuscany Region n. 677 of 8.4.2014.

The aim of this project is to analyze the potential contribution of IGRA test, QuantiFERON-TB Gold In Tube test (QTF-GIT, Cellestis Limited, Carnegie, Victoria, Australia) in the diagnosis of tuberculosis (TB - active or latent) in pediatric subjects aged between 0 and 17 years recently exposed to infection (indicated as "contacts") or with clinical suspicion of active TB, and to compare the results obtained with those of the TuberculinSkin Test (TST), which is the gold standard. The research project is expected to enroll up to 50 pediatric patients (0- 17 years) over a 4-year study. Children with access to Ambulatory structures or hospitalized at University Infectious Diseases Clinic or Pediatric Clinic, University Hospital of Siena, or with access to Ambulatory or hospitalized at Pediatric Clinic USL 9 Grosseto will be enrolled. Once obtained the informed consent of patients' parents or legal guardians, patients will be enrolled. The doctor will administer a clinical-anamnestic questionnaire (CRF), relative to the country of birth and residence, date of arrival in Italy and any stays in the country of origin (in case of foreign patient), travels abroad, risk factors for infectious diseases, type of contact with any index case, previous vaccination with BCG, date and outcome of the TST, clinical symptoms and signs suggestive of active TB, report of any instrumental investigation. Together with the collection of blood samples for routine purposes, an additional blood sample will be taken so to run experimental IGRA test. Also patients for whom their medical doctor will independently order to run QTF-GIT test as necessary tool for the clinical diagnosis of TB will be included in the study.

A retrospective analysis will be performed on patient pertaining to participant Clinics, from 1 January 2012 to 31 May 2015. Such analysis will be performed on those patients for which their medical doctor requested both intradermal Mantoux and IGRA test.

Main objectives:

1. Estimation of concordance between QuantiFERON-TB Gold In Tube and TST in pediatric patients exposed to TB
2. Evaluation of the sensitivity of the test QTF-GIT in patients with active tuberculosis disease
3. Evaluation of specificity of test QTF-GIT in not infected patients

Secondary objectives:

* Evaluation of the possible use of QTF-GIT, together with TST, to improve the diagnosis of latent or active tuberculosis infection in pediatric subjects.
* Evaluation of the possible diagnostic use of QTF-GIT in the child, with special attention to children <5 years.

ELIGIBILITY:
Inclusion Criteria:

* Age between 0 to 17 years
* Willingness to provide informed consent (parents or legal guardians)
* Contact with TB case and/or clinical suspect of active TB

Exclusion Criteria:

* Acquired or congenital immune deficiencies
* Oncohematologic diseases

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study will be performed on children hospitalized at Policlinico Santa Maria alle Scotte (Infectious Dieseases and Pediatrics wards), at Pediatric Clinic of Grosseto USL9, and from the ambulatories of the above mentioned hospitals.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-04; Primary Completion 2019-04 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with concordance of QTF-GIT test and TST,among children exposed to TB | up to 4 years
Number of patients with positivity of QTF-GIT in comparison with TST among children with active tuberculosis disease | up to 4 years
Number of patients with a negative QTF-GIT test in comparison of TST, among non-infected children | up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Montagnani, PhD, MD, Principal Investigator — Università di Siena - Azienda Ospedaliera Santa Maria alle Scotte
Locations (3):
- Italy (3):
  - UOC Pediatria, USL9, Grosseto, Grosseto, GR
  - UOC Pediatria c/o Policlinico Le Scotte, Viale Mario Bracci 16, Siena, SI
  - UOC Malattie Infettive Universitarie c/o Policlinico Le Scotte, Viale Mario Bracci 16, Siena

REFERENCES:
- [Result] Huebner RE, Schein MF, Bass JB Jr. The tuberculin skin test. Clin Infect Dis. 1993 Dec;17(6):968-75. doi: 10.1093/clinids/17.6.968. No abstract available. PMID 8110954
- [Result] Andersen P, Munk ME, Pollock JM, Doherty TM. Specific immune-based diagnosis of tuberculosis. Lancet. 2000 Sep 23;356(9235):1099-104. doi: 10.1016/s0140-6736(00)02742-2. PMID 11009160
- [Result] Munoz L, Santin M. Interferon-gamma release assays versus tuberculin skin test for targeting people for tuberculosis preventive treatment: an evidence-based review. J Infect. 2013 Apr;66(4):381-7. doi: 10.1016/j.jinf.2012.12.005. Epub 2013 Jan 5. PMID 23298892
- [Result] Diel R, Goletti D, Ferrara G, Bothamley G, Cirillo D, Kampmann B, Lange C, Losi M, Markova R, Migliori GB, Nienhaus A, Ruhwald M, Wagner D, Zellweger JP, Huitric E, Sandgren A, Manissero D. Interferon-gamma release assays for the diagnosis of latent Mycobacterium tuberculosis infection: a systematic review and meta-analysis. Eur Respir J. 2011 Jan;37(1):88-99. doi: 10.1183/09031936.00115110. Epub 2010 Oct 28. PMID 21030451
- [Result] Chiappini E, Accetta G, Bonsignori F, Boddi V, Galli L, Biggeri A, De Martino M. Interferon-gamma release assays for the diagnosis of Mycobacterium tuberculosis infection in children: a systematic review and meta-analysis. Int J Immunopathol Pharmacol. 2012 Jul-Sep;25(3):557-64. doi: 10.1177/039463201202500301. PMID 23058005
- [Result] Sollai S, Galli L, de Martino M, Chiappini E. Systematic review and meta-analysis on the utility of Interferon-gamma release assays for the diagnosis of Mycobacterium tuberculosis infection in children: a 2013 update. BMC Infect Dis. 2014;14 Suppl 1(Suppl 1):S6. doi: 10.1186/1471-2334-14-S1-S6. Epub 2014 Jan 8. PMID 24564486
- [Result] Blandinieres A, de Lauzanne A, Guerin-El Khourouj V, Gourgouillon N, See H, Pedron B, Faye A, Sterkers G. QuantiFERON to diagnose infection by Mycobacterium tuberculosis: performance in infants and older children. J Infect. 2013 Nov;67(5):391-8. doi: 10.1016/j.jinf.2013.06.011. Epub 2013 Jun 22. PMID 23796868
- [Result] Marais BJ, Gie RP, Schaaf HS, Hesseling AC, Obihara CC, Starke JJ, Enarson DA, Donald PR, Beyers N. The natural history of childhood intra-thoracic tuberculosis: a critical review of literature from the pre-chemotherapy era. Int J Tuberc Lung Dis. 2004 Apr;8(4):392-402. PMID 15141729